CLINICAL TRIAL: NCT04079023
Title: Prospective Pathophysiological Evaluation of Alcohol Intake and Metabolism After Sleeve Gastrectomy
Brief Title: Alcohol Metabolism After Sleeve Gastrectomy
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Collaborators: Azienda vinicola Casal del Giglio (Unknown)
Responsible Party: Principal Investigator, Angelo Iossa, principal investigator, University of Roma La Sapienza
Other Study IDs: Lasapienza2019
Record Dates: First submitted 2019-08-29; First posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Alcohol Metabolism Modifier Adverse Reaction; Bariatric Surgery Candidate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Obese: 30 obese patients (12 M/ 18 F) with a mean BMI of 46 candidate to SG Alcohol drink mean volume: 158 Ml administered in 10 minutes
  Interventions: Procedure: Sleeve Gastrectomy

INTERVENTIONS:
Procedure: Sleeve Gastrectomy — Subtotal vertical gastrectomy

SUMMARY:
This prospective study aimed to determine the alcohol intake symptoms and alcohol metabolism before and 12 months after sleeve gastrectomy (SG) by evaluating blood alcohol content (BAC) and urinary alcohol metabolite levels against the amount of alcohol consumed to reveal the occurrence of any AUD..

DETAILED DESCRIPTION:
The sample size was selected based on the number of obese patients who underwent SG at our Bariatric Center of Excellence IFSO-EC over the last 12 months, and the end-time of evaluation was estimated independently due to the lack of high evidence-based studies, such as randomized trials or meta-analyses, focusing on the impact of alcohol on the bariatric population. Considering the requirement of 200 patients to obtain a 95% confidence level, a sample size of 30 patients was selected to achieve a confidence interval (margin of error) of 16.54. Data were collected and analyzed as mean and standard deviation.

Inclusion criteria were patients aged 21-60 years with BMI of 35-49 kg/m2 who were planned to undergo primary SG and agreed to participate in the study and undergo evaluation before and after SG. Exclusion criteria were non-drinker, previous history of alcoholism, T2D diagnosed based on the ADA criteria for diabetes 2016, hepatic cirrhosis, nonalcoholic steatohepatitis or hepatitis C/cirrhosis, previous resective gastrointestinal surgery (elective or emergent), previous bariatric procedures, and cholelithiasis (symptomatic or asymptomatic).

The amount of wine to be consumed was calculated based on the patient's total water body mass at the time of measurement (0-6-12 months) because alcohol is distributed throughout the entire water body mass without adhering to plasma proteins and its solubility in fat and bones is undetectable. The amount of wine (mL) was calculated using the following formula reported by Maluenda et al.: 3.6 × total body water (TBW). Body mass composition was measured using BIA 101 ASE (Akern SRL, Firenze, Italy) after 2-h fasting and emptying the bladder and analyzed using the Bodygram Plus software V.1.0 (Akern SRL, Firenze, Italy). The red wine Madreselva containing 14% of alcohol per liter, which is certified for standard alcohol level at packaging and durability of over 3 years, was kindly provided by the local factory Casal del Giglio. At time 0, BAC was measured using an ethanol assay kit (DiaSys Diagnostic Systems GmbH) at 15, 30, and 60 mins and then every 30 min after alcohol intake until the ethanol level of 0 g/L was obtained. Six hours of fasting before and after wine consumption were observed. Blood examination was repeated at 6 and 12 months after SG. At time 0 and 12 months after SG, the urinary metabolite (ethanol and acetaldehyde) levels were evaluated after urinary bladder filling for 2 h and the liver function [albumin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma-glutamyl transferase (GGT), bilirubin, lactate dehydrogenase (LD), alkaline phosphatase (ALP), uric acid, and INR] was evaluated to detect alcohol-induced changes. Each patient's subjective attitude to alcohol consumption was evaluated at 0- and 12-months using alcohol use disorder identification test (AUDIT); score ≥ 8 was considered to indicate alcohol dependence and those patients were excluded as per the study criteria. The perception of symptoms, including the most common symptoms of alcoholization (euphoria and diaphoresis) and intoxication (anxiety, nausea/vomiting, and flushing), after alcohol consumption was evaluated using a newly developed symptom alcoholization post obesity surgery (SAPoS) scoring system (not validated). This scoring system was created based on the experience gained during clinical check-ups and investigates the symptoms occurring after alcohol consumption. The data on BAC at 0-6-12 months, urinary metabolite levels at 0-12 months, and SAPoS scores at 0-6-12 months were compared. Differences were considered statistically significant at p < 0.05

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21 ≤ 60 years
* BMI ≥ 35 ≤49 Kg/m2
* Candidate to LSG
* Accepts to scheduled follow-up scheme

Exclusion Criteria:

* Non-drinker
* Previous history of alcoholism
* DMTII
* Hepatic cirrhosis, Nonalcoholic steatohepatitis (NASH) or HCV hepatitis/cirrhosis
* Previous resective gastro-intestinal surgery
* Cholelithiasis

Ages: 21 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Obese, normal drinker
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
blood alcohol content (BAC) | 0, 6 and 12 months
  Change in BAC after SG
urinary alcohol metabolite | 0 and 12 Months
  change in alcohol metabolite (ethanol and acetaldehyde) after SG

SECONDARY OUTCOMES:
alcohol addiction | 0, 6 and 12 Months
  change in alcohol preferences measured with AUDIT( Alcol Use disorders Identification TesT) test

CONTACTS AND LOCATIONS:
Overall Officials: Angelo A Iossa, Principal Investigator — University of Roma La Sapienza
Locations (1):
- University of Rome "la sapienza", Latina, Italy

IPD SHARING:
Plan to Share IPD: No